CLINICAL TRIAL: NCT03081429
Title: A Prospective Cohort Study of Perioperative Covert Stroke and Postoperative Cognitive Dysfunction in Elderly Patients Undergoing Noncardiac Surgery
Brief Title: A Prospective Cohort Study of Perioperative Covert Stroke and Postoperative Cognitive Dysfunction
Acronym: PRECISION
Status: Completed | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Yuming Peng, Professor, Beijing Tiantan Hospital
Other Study IDs: 2017-3-10
Record Dates: First submitted 2017-03-10; First posted 2017-03-16 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Anesthesia; Covert Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With stroke
- Without stroke

SUMMARY:
With the development of population aging, the incidence of covert stroke gradually increased. Currently, there is still lack of prospective cohort study with large sample size on the relationship between perioperative covert stroke and postoperative cognitive outcomes. The investigators will perform a prospective cohort study. The aim of the study is to determine whether there is an association between perioperative covert stroke and postoperative cognitive outcomes in elderly patients undergoing noncardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Eligible patients were aged ≥60 years and scheduled for elective non-cardiac surgery with general anesthesia, with or without concomitant regional analgesia. They were expected to have surgery lasting at least 2 hours of anesthesia and to stay in the hospital at least 2 days thereafter.

Exclusion Criteria:

* Patients have MRI contraindications, cannot complete the cognitive evaluation, undergo carotid artery surgery or refuse to sign informed consent will be excluded from the trial.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population will be selected from patients who schedule to receive elective noncardiac surgery in Beijing Tiantan Hospital and Chinese People's Liberation Army General Hospital.
Sampling Method: Probability Sample
Enrollment: 934 (Actual)
Dates: Start 2018-05-23 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
The incidence of perioperative stroke | Postoperative 1-7 days
  Stroke is diagnosed by MRI

SECONDARY OUTCOMES:
Postoperative cognitive function | 1 day before surgery; and 7 days, 3 months, 1 year after surgery
  Cognitive assessment will be conducted by trained research members who are blinded to the clinical diagnosis, treatment and MRI. The Mini-mental State Examination, Montreal cognitive assessment-basic, Mini-Mental State Examination telephone scales, Montreal Cognitive Assessment telephone scales, and Telephone Interview of Cognitive Status scale will be used to assess the cognitive function. Postoperative cognitive dysfunction is defined as at least 2 standard deviation reduction on the Mini-Mental State Examination telephone scales or Montreal Cognitive Assessment telephone scales or a Telephone Interview of Cognitive Status scale scores≤27.
Postoperative delirium | twice a day (from 8:00 to 10:00 and from 18:00 to 20:00) during the first postoperative 5 days
  The Confusion Assessment Method for the Intensive Care Unit scale (CAM-ICU) or 3 min diagnostic interview for CAM (3D-CAM) will be applied to assess delirium.
Recovery quality | 1 day before surgery; and 7 days, 30 days, 3 months after surgery
  The Modified Rankin Scale (mRS) and Lawton instrumental activities of daily living scale (IADL) will be applied to assess the recovery quality.
The quality of life | 1 day before surgery; and 7 days, 30 days, 3 months after surgery
  The quality of life will be assessed with the EuroQol-5D (EQ-5D) scale.
Depression state | 1 day before surgery; and 7 days, 30 days, 3 months after surgery
  Depression state will be assessed with the Geriatric Depression Scale, Generalized Anxiety Disorder-7 and Patient Health Questionnaire-9.
The incidence of comorbidity. | 30 days and 3 months after surgery
  The incidence of myocardial infarction, cardiac arrest, pulmonary embolism, sepsis, surgical site infection and persistent postoperative pain.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Beijing TianTan Hospital, Beijing
  - Chinese People's Liberation Army General Hospital, Beijing

REFERENCES:
- [Derived] Cui Q, Wang D, Zeng M, Dong J, Jin H, Hu Z, Zhang Y, Peng Y, Han R. Association of postoperative covert stroke and cognitive dysfunction among elderly patients undergoing non-cardiac surgery: protocol for a prospective cohort study (PRECISION study). BMJ Open. 2020 Jan 6;10(1):e034657. doi: 10.1136/bmjopen-2019-034657. PMID 31911527